CLINICAL TRIAL: NCT01318902
Title: An Open-Label, Dose-Escalation, Phase 1 Study of the Oral Formulation of MLN9708 Administered Weekly in Adult Patients With Relapsed or Refractory Light-Chain (AL) Amyloidosis Who Require Further Treatment
Brief Title: Study of Oral Ixazomib in Adult Participants With Relapsed or Refractory Light Chain Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16007; 2010-022497-13 (EudraCT Number); U1111-1168-1192 (Registry Identifier: WHO (UTN ))
Record Dates: First submitted 2011-03-15; First posted 2011-03-21 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Light-Chain Amyloidosis
Keywords: Drug therapy
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — ixazomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Escalation Cohort: Ixazomib 4.0 mg (Experimental): Ixazomib 4.0 mg, capsule, orally, once weekly on Days 1, 8 and 15 during each 28-day treatment cycle for 3 cycles. If there was no hematologic response, dexamethasone 40 mg, tablet, orally was added once on Days 1 to 4 of every cycle, beginning in Cycle 4 for 3 additional cycles. If there was no hematologic response the participant was discontinued. Participants with hematologic response continued treatment up to maximum 12 cycles.
  Interventions: Drug: Ixazomib; Drug: Dexamethasone
- Dose Escalation Cohort: Ixazomib 5.5 mg (Experimental): Ixazomib 5.5 mg, capsule, orally, once weekly on Days 1, 8 and 15 during each 28-day treatment cycle for 3 cycles. If there was no hematologic response, dexamethasone 40 mg, tablet, orally was added once on Days 1 to 4 of every cycle, beginning in Cycle 4 for 3 additional cycles. If there was no hematologic response the participant was discontinued. Participants with hematologic response continued treatment up to maximum 12 cycles.
  Interventions: Drug: Ixazomib; Drug: Dexamethasone
- Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) (Experimental): Ixazomib 4.0 mg, capsule, orally, on Days 1, 8 and 15 during a 28-day treatment cycle until progressive disease (PD) or unacceptable toxicity, for participants with relapsed or refractory amyloidosis and who were not treated with any other proteasome inhibitor (PI). Duration of treatment was up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months.
  Interventions: Drug: Ixazomib
- Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed) (Experimental): Ixazomib 4.0 mg, capsule, orally, on Days 1, 8 and 15 during a 28-day treatment cycle until PD or unacceptable toxicity, for participants with relapsed or refractory amyloidosis and who were previously treated with any other PI. Duration of treatment was up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules.
  Other Names: MLN9708
Drug: Dexamethasone — Dexamethasone tablets.
  Arms: Dose Escalation Cohort: Ixazomib 4.0 mg; Dose Escalation Cohort: Ixazomib 5.5 mg

SUMMARY:
This study will include participants with previously treated systemic relapsed or refractory light-chain (AL) amyloidosis who require further therapy and will be aimed at determining the safety profile and the maximum tolerated dose/recommended phase 2 dose of MLN9078 (Ixazomib) administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older
* Biopsy-proven systemic relapsed or refractory light-chain (AL) amyloidosis, which after at least 1 prior therapy, in the investigator's opinion, requires further treatment
* If received stem cell transplant, must be at least 3 months posttransplantation and recovered from side effects
* Must have measurable disease defined as serum differential free light chain concentration ≥ 40 mg/L
* Must have objective measurable organ (heart or kidney) amyloid involvement
* Must have cardiac biomarker risk stage I or II disease
* Must have adequate hematologic, hepatic, and renal function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Female participants who are postmenopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to abstain from heterosexual intercourse
* Male participants who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Voluntary written consent

Exclusion Criteria

* Peripheral neuropathy that is greater or equal to Grade 2
* Cardiac status as described in protocol
* Severe diarrhea (≥ Grade 3) not controllable with medication or requires administration of total parenteral nutrition
* Known gastrointestinal condition or procedure that could interfere with swallowing or the oral absorption of tolerance of MLN9708
* Uncontrolled infection requiring systematic antibiotics
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Presence of other active malignancy with the exception of nonmelanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate-specific antigen is within normal limit, or any completely resected carcinoma in situ
* Female participants who are lactating or pregnant
* Major surgery within 14 days before the first dose of study drug
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (10):
- United States (6):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- University Health Network, Toronto, Ontario, Canada
- CHU Limoges, Department of Hematology and Cell Therapy, Reference Center for AL amyloidosis, Limoges, France
- Universitatsklinikum Heidelberg Innere Medizin V; Hamatologie, Onkologie und Rheumatologie, Heidelberg, Germany
- Amyloidosis Research & Treatment Center, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Result] Sanchorawala V, Comenzo R, Zonder J, Kukreti V, Cohen A, Dispenzieri A, et al. MLN9708, an investigational oral proteasome inhibitor (PI), in relapsed or refractory lightchain (AL) amyloidosis. Clinical Lymphoma Myeloma and Leukemia 2013;13(suppl 1):S153-4; abstr P-229.
- [Result] Sanchorawala V, Zonder J, Comenzo R, Schönland S, Dispenzieri A, Berg D, et al. Poster Presentation: Phase 1 study of MLN9708, a novel, investigational oral proteasome inhibitor, in patients with relapsed or refractory light-chain amyloidosis. XIII International Symposium on Amyloidosis, Groningen, The Netherlands 2012.
- [Result] Merlini G, Sanchorawala V, Zonder J, Kukreti V, Schonland S, Jaccard A, et al. MLN9708, a novel, investigational oral proteasome inhibitor, in patients with relapsed or refractory light-chain amyloidosis (AL): results of a phase 1 study. In: 54th ASH Annual Meeting and Exposition; 2012 8-11 December; Atlanta, GA; p. abstr 731.
- [Derived] Sanchorawala V, Palladini G, Kukreti V, Zonder JA, Cohen AD, Seldin DC, Dispenzieri A, Jaccard A, Schonland SO, Berg D, Yang H, Gupta N, Hui AM, Comenzo RL, Merlini G. A phase 1/2 study of the oral proteasome inhibitor ixazomib in relapsed or refractory AL amyloidosis. Blood. 2017 Aug 3;130(5):597-605. doi: 10.1182/blood-2017-03-771220. Epub 2017 May 26. PMID 28550039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in the United States, Canada, France, Germany and Italy from 27 April 2011 to 13 November 2018.
Pre-assignment Details: Participants with previously treated systemic light chain (AL) amyloidosis were enrolled in 2 dose escalation cohorts and were treated with ixazomib 4.0 or 5.5 mg. Participants with relapsed or refractory amyloidosis were enrolled in 2 dose expansion cohorts and treated with ixazomib 4.0 mg in proteosome inhibitor (PI) Naive and PI Exposed groups.
Period: Overall Study
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Started | 6 | 5 | 5 | 11
Completed (Completed=participants who completed maximum cycles per protocol and who had progressive disease.) | 5 | 2 | 3 | 5
Not Completed | 1 | 3 | 2 | 6
Not completed — Symptomatic Deterioration | 0 | 1 | 1 | 2
Not completed — Withdrawal by Patient | 0 | 1 | 0 | 3
Not completed — Unsatisfactory Therapeutic Response | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Terminated by Sponsor | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed) | Total
Number analyzed (Participants) | 6 | 5 | 5 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6.15) | 69.0 (8.51) | 65.8 (6.26) | 66.7 (8.49) | 66.2 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 5 | 13
  Male | 4 | 1 | 3 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 5 | 8 | 22
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 5 | 3 | 10 | 23
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 1
  Not Reported | 0 | 0 | 0 | 1 | 1
  Other | 1 | 0 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 173.26 (7.504) | 159.17 (11.043) | 173.56 (20.728) | 167.35 (9.056) | 168.30 (12.436)
Weight [Mean (Standard Deviation); unit: kg] | 76.78 (5.464) | 64.03 (12.664) | 85.83 (40.280) | 70.96 (11.402) | 73.73 (19.536)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy.
Time Frame: From the first dose of study drug plus 30 days after last dose of study drug or until the initiation of subsequent antineoplastic therapy (Up to approximately 13 months)
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 5 | 5 | 11
Participants
  TEAE | 6 | 5 | 5 | 10
  SAE | 3 | 5 | 5 | 5

2. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values Reported as TEAE
Description: The number of participants with any clinically significant abnormal standard safety laboratory values collected throughout the study reported as TEAEs. Parameters assessed were hematology, serum chemistry and urinalysis. Abnormal laboratory values were assessed as an AE if that value leads to discontinuation or delay in treatment, dose modification, therapeutic intervention, or is considered by the investigator to be a clinically significant change from baseline.
Time Frame: as for outcome 1
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 5 | 5 | 11
Participants
  Thrombocytopenia | 2 | 0 | 2 | 2
  Anaemia | 2 | 0 | 2 | 0
  Neutropenia | 0 | 0 | 0 | 1
  Hyponatraemia | 1 | 0 | 1 | 1
  Hypokalaemia | 1 | 0 | 0 | 1
  Blood creatinine increased | 1 | 0 | 0 | 1
  Platelet count decreased | 0 | 2 | 0 | 0

3. Primary Outcome: Number of Participants With Peripheral Neuropathy Reported as a TEAE
Description: Neurotoxicity was assessed as the number of participants with the TEAE of peripheral neuropathy.
Time Frame: as for outcome 1
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 5 | 5 | 11
Participants
  Peripheral sensory neuropathy | 1 | 0 | 1 | 1
  Neuropathy peripheral | 1 | 0 | 0 | 0

4. Primary Outcome: Maximum Tolerated Dose (MTD) of Ixazomib
Description: MTD was highest dose of Ixazomib, at which <=1 of 6 participants experienced dose-limiting toxicity (DLT). DLT was defined using National Cancer Institute Common Terminology Criteria for Adverse Events, v 4.03 as: Grade 4 neutropenia (absolute neutrophil count <500 cells/mm^3) for >7 days;Grade 3 neutropenia with fever or infection;Grade 4 thrombocytopenia (platelets < 25,000/mm^3) for >7 days;Grade 3 thrombocytopenia with clinically significant bleeding;platelet count <10,000/mm^3;Grade 2 peripheral neuropathy with pain or >=Grade 3 peripheral neuropathy; >=Grade 3 nausea/emesis, diarrhea controlled by supportive therapy;Grade 3 QTc prolongation (QTc >500 msec);any >=Grade 3 nonhematologic toxicity except Grade 3 arthralgia/myalgia;or <1 week Grade 3 fatigue;delay in initiation of the subsequent therapy cycle by >2 weeks;other >=Grade 2 study drug-related nonhematologic toxicities requiring therapy discontinuation, considered possibly related to therapy as assessed by Investigator.
Time Frame: Cycle 1 (28 days)
Population: DLT-evaluable population included all participants who received all Cycle 1 doses of ixazomib or experienced a DLT in Cycle 1.
Measure: Number; unit: mg
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg
Number analyzed (Participants) | 6 | 5
mg | 4 | 4

5. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Ixazomib
Description: The RP2D is the maximum tolerated dose (MTD) or less. The MTD is defined as the dose range at which ≤ 1 of 6 evaluable participants experience dose limiting toxicities (DLT) within the first 28 days of treatment (end of Cycle 1). The RP2D of Ixazomib was determined in dose escalation group on the basis of the totality of safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) data observed in Cycle 1.
Time Frame: Cycle 1 (28 days)
Population: as for outcome 4
Measure: Number; unit: mg
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg
Number analyzed (Participants) | 6 | 5
mg | 4 | 4

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Cycle 1: Day 1 (MTD cohort participants only, 4.0 mg) and Day 15 (all participants enrolled in the study): predose (within 1 hour (hr) before dosing), and postdose at multiple timepoints up to 168 hr
Population: Pharmacokinetic (PK) analysis population included all participants who received at least 1 dose of ixazomib and had sufficient ixazomib concentration-time data and dosing data to permit calculation of ixazomib plasma PK parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Ixazomib 4.0 mg: Ixazomib 4.0 mg, capsule, orally, once weekly on Days 1 and 15 during each 28-day treatment cycle for all the participants from dose escalation and expansion cohorts were evaluated in this arm group. Duration of treatment was up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months.
- Ixazomib 5.5 mg: Ixazomib 5.5 mg, capsule, orally, once weekly on Days 1, 8 and 15 during each 28-day treatment cycle for 3 cycles. If there was no hematologic response, dexamethasone was added on Days 1 to 4 of every cycle, beginning in Cycle 4 for 3 additional cycles. The maximum duration of treatment was up to 12 cycles.
Arm/Group | Ixazomib 4.0 mg | Ixazomib 5.5 mg
Number analyzed (Participants) | 20 | 2
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 15 | 0
  Cycle 1, Day 1 | 54.00 [16.7 to 163.0] |
  Cycle 1, Day 15: number analyzed (Participants) | 18 | 2
  Cycle 1, Day 15 | 51.26 [10.7 to 131.0] | 92.20 [61.4 to 123.0]

7. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Ixazomib
Time Frame: as for outcome 6
Population: PK analysis population included all participants who received at least 1 dose of ixazomib and had sufficient ixazomib concentration-time data and dosing data to permit calculation of ixazomib plasma PK parameters. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | Ixazomib 4.0 mg | Ixazomib 5.5 mg
Number analyzed (Participants) | 20 | 2
hours
  Cycle 1, Day 1: number analyzed (Participants) | 15 | 0
  Cycle 1, Day 1 | 1.0000 [0.500 to 2.000] |
  Cycle 1, Day 15: number analyzed (Participants) | 18 | 2
  Cycle 1, Day 15 | 1.0000 [0.500 to 6.080] | 0.7500 [0.500 to 1.000]

8. Secondary Outcome: Ctrough: Plasma Concentration Immediately Prior to Dosing for Ixazomib
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Ixazomib 4.0 mg | Ixazomib 5.5 mg
Number analyzed (Participants) | 20 | 2
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 15 | 0
  Cycle 1, Day 1 | 2.1539 [0.000 to 14.400] |
  Cycle 1, Day 15: number analyzed (Participants) | 15 | 2
  Cycle 1, Day 15 | 2.9140 [1.010 to 6.750] | 5.3300 [4.410 to 6.250]

9. Secondary Outcome: AUC0-168: Area Under the Plasma Concentration-time Curve From Time 0 to 168 Hours Post-dose for Ixazomib
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Full Range); unit: hr*ng/mL
Arm/Group | Ixazomib 4.0 mg | Ixazomib 5.5 mg
Number analyzed (Participants) | 20 | 2
hr*ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 14 | 0
  Cycle 1, Day 1 | 861.0 [237 to 5010] |
  Cycle 1, Day 15: number analyzed (Participants) | 15 | 2
  Cycle 1, Day 15 | 1078.1 [465 to 2220] | 1725.0 [1240 to 2210]

10. Secondary Outcome: Emax: Maximum Observed Percent Inhibition of Whole Blood 20S Proteasome
Time Frame: as for outcome 6
Population: Pharmacodynamic (PD) analysis population: all participants who received at least 1 dose of ixazomib and had whole blood 20S proteasome inhibition-time data and dosing data to permit calculation of PD parameters. Data was only collected for ixazomib 4.0 mg arm group. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Ixazomib 4.0 mg
Number analyzed (Participants) | 15
percentage of inhibition
  Cycle 1, Day 1 | 54.10 (12.438)
  Cycle 1, Day 15: number analyzed (Participants) | 13
  Cycle 1, Day 15 | 61.09 (11.846)

11. Secondary Outcome: TEmax: Time to Maximum Observed Effect (Emax) of Whole Blood 20S Proteasome Inhibition for Ixazomib
Time Frame: as for outcome 6
Population: PD analysis population: all participants who received at least 1 dose of ixazomib and had whole blood 20S proteasome inhibition-time data and dosing data to permit calculation of PD parameters. Data was only collected for ixazomib 4.0 mg arm group. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | Ixazomib 4.0 mg
Number analyzed (Participants) | 15
hours
  Cycle 1, Day 1 | 1.0000 [0.500 to 6.000]
  Cycle 1, Day 15 | 1.0300 [0.500 to 6.020]

12. Secondary Outcome: AUE0-168: Area Under Effect Curve of Whole Blood 20S Proteasome Inhibition From Zero to Concentration at 168 Hours for Ixazomib
Time Frame: as for outcome 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr*percentage of inhibition
Arm/Group | Ixazomib 4.0 mg
Number analyzed (Participants) | 15
hr*percentage of inhibition
  Cycle 1, Day 1: number analyzed (Participants) | 14
  Cycle 1, Day 1 | 3333.6 (1377.24)
  Cycle 1, Day 15: number analyzed (Participants) | 10
  Cycle 1, Day 15 | 3943.0 (2322.96)

13. Secondary Outcome: Number of Participants With Best Organ Response to Treatment Based on Investigators Assessment
Description: Organ response rate was estimated as the number of participants with documented organ response (ie. Heart or kidney ). Treatment response of amyloid-related organs were identified based on national cancer institute, common terminology criteria for adverse events (NCI CTCAE) Version 4.02 criteria.
Time Frame: At Cycles 3, 6, 9, and 12; every 6 months thereafter until disease progression or the initiation of subsequent antineoplastic therapy and at end of treatment (EOT) visit (Up to approximately 12 months)
Population: Organ response-evaluable population included all participants who received at least 1 cycle of ixazomib, had amyloid involvement of at least kidney or heart at baseline, and had at least 1 postbaseline organ response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 2 | 4 | 8
Participants | 2 | 0 | 2 | 2

14. Secondary Outcome: Number of Participants With Best Hematologic Response to Treatment Based on Investigators Assessment
Description: The overall hematologic response rate is defined as number of participants with complete response (CR) or partial response (PR) or very good partial response (VGPR) as assessed by the investigator. Response is determined according to standardized criteria using a central laboratory. CR=serum and urine negative for monoclonal protein by immunofixation; or free light chain ratio normal; < 5% plasma cells in bone marrow without clonal dominance. PR=reduction in dFLC > 50%. VGPR= dFLC < 40 mg/L.
Time Frame: Day 22 to 28 in each cycle and end of treatment visit; then every 6 weeks thereafter until disease progression or initiation of subsequent antineoplastic therapy (Up to approximately 12 months)
Population: Hematologic response-evaluable population included all participants who received at least 1 cycle of ixazomib, had measureable disease at baseline, and had at least 1 postbaseline hematologic response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 3 | 4 | 11
Participants | 4 | 0 | 4 | 3

15. Secondary Outcome: Time to First Hematologic Response
Description: Time to first hematologic response, measured as the time from the first dose of ixazomib to the date of first documentation of a hematologic response.
Time Frame: From the date of the first dose of ixazomib to the date of first documentation of a hematologic response (Up to approximately 12 months)
Population: Hematologic response-evaluable population: all participants who received at least 1 cycle of ixazomib, had measureable disease at baseline, had >=1 postbaseline hematologic response. No participants had hematologic response for ixazomib 5.5 mg arm group thus were not analyzed. Data is reported for participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 4 | 0 | 4 | 3
months | 0.79 [0.7 to 1.8] |  | 3.45 [0.9 to 4.4] | 2.11 [1.0 to 3.7]

16. Secondary Outcome: Time to First Organ Response
Description: Time to first organ response, measured as the time from the first dose of ixazomib to the date of first documentation of a organ response.
Time Frame: From the date of the first dose of ixazomib to the date of first documentation of a organ response (Up to approximately 12 months)
Population: Organ Response-Evaluable population included participants who received at least 1 cycle of ixazomib, who had amyloid involvement of at least kidney or heart at baseline, and who had at least 1 postbaseline organ response assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 2 | 0 | 2 | 2
months | 6.85 [2.7 to 11] |  | 9.55 [2.7 to 16.4] | 6.85 [2.5 to 11.2]

17. Secondary Outcome: Duration of Hematologic Response
Description: Duration of hematologic response, measured as the time from the date of first documentation of a hematologic response to the date of hematologic disease progression.
Time Frame: From the date of first documentation of a hematologic response to the date of hematologic disease progression (Up to approximately 12 months)
Population: as for outcome 15
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 4 | 0 | 4 | 3
months | 12.9 [7.4 to 16.1] |  | 69.5 [7.8 to 75.2] | 19.7 [0.4 to 33.2]

18. Secondary Outcome: Duration of Organ Response
Description: Duration of organ response, measured as the time from the date of first documentation of a organ response to the date of organ disease progression.
Time Frame: From the date of first documentation of a organ response to the date of organ disease progression (Up to approximately 12 months)
Population: Organ Response-Evaluable population included participants who received at least 1 cycle of ixazomib, who had amyloid involvement of at least kidney or heart at baseline, and who had at least 1 postbaseline organ response assessment. Number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 2 | 0 | 1 | 2
months | 4.1 [0 to 8.2] |  | 20.5 [20.5 to 20.5] | 18.25 [0 to 36.5]

19. Secondary Outcome: Time to Hematologic Disease Progression
Description: Time to hematologic progression, measured as the time from the date of the first dose of ixazomib to the date of first documented hematologic disease progression.
Time Frame: From the date of the first dose of ixazomib to the date of first documented hematologic disease progression (Up to approximately 12 months)
Population: Safety population included all participants who received at least 1 dose of ixazomib. Data is reported for participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 4 | 1 | 2 | 5
months | 14.8 [1.6 to 17.0] | NA [NA to NA] — Median, lower and upper limit was not estimable due to low number of participants with events. | 73.0 [0.0 to 78.7] | 8.3 [0.9 to 36.8]

20. Secondary Outcome: Time to Organ Disease Progression
Description: Time to organ disease progression, measured as the time from the date of the first dose of ixazomib to the date of first documented organ disease progression.
Time Frame: From the date of the first dose of ixazomib to the date of first documented organ disease progression (Up to approximately 12 months)
Population: as for outcome 16
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 2 | 0 | 2 | 2
months | 11 [11 to 11] |  | 12.85 [2.5 to 23.2] | 25.15 [2.5 to 47.8]

21. Secondary Outcome: Hematologic Disease Progression-Free Survival (PFS)
Description: Hematologic disease PFS, measured as the time from the date of the first dose of ixazomib to the date of hematologic disease progression or death.
Time Frame: From the date of the first dose of ixazomib to the date of hematologic disease progression or death (Up to approximately 12 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 4 | 3 | 3 | 6
months | 14.8 [1.6 to 17.0] | 7.2 [0.0 to 9.2] | 73.0 [0.6 to 78.7] | 8.3 [0.9 to 36.8]

22. Secondary Outcome: Organ Disease Progression-Free Survival (PFS)
Description: Organ disease PFS, measured as the time from the date of the first dose of ixazomib to the date of organ disease progression or death.
Time Frame: From the date of the first dose of ixazomib to the date of organ disease progression or death (Up to approximately 12 months)
Population: as for outcome 16
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 2 | 4 | 8
months | NA [NA to NA] — Data was not estimable due to low number of participants with events. | NA [NA to NA] — Data was not estimable due to low number of participants with events. | NA [NA to NA] — Data was not estimable due to low number of participants with events. | NA [NA to NA] — Data was not estimable due to low number of participants with events.

23. Secondary Outcome: Percentage of Participants With One Year Hematologic Disease PFS
Description: One-year survival, defined as the patient survival probability at 1 year after the date of first dose of ixazomib.
Time Frame: From the date of the first dose of ixazomib to the date of hematologic disease progression or death (Up to 1 year)
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
Number analyzed (Participants) | 6 | 0 | 5 | 11
percentage of participants | 83.3 |  | 80.0 | 21.5

ADVERSE EVENTS:
Time Frame: From the first dose of study drug plus 30 days after last dose of study drug or until the initiation of subsequent antineoplastic therapy (Up to approximately 13 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation Cohort: Ixazomib 4.0 mg | Dose Escalation Cohort: Ixazomib 5.5 mg | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 1/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/5 | 5/5 | 5/11
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 5/5 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort: Ixazomib 4.0 mg (N=6) | Dose Escalation Cohort: Ixazomib 5.5 mg (N=5) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) (N=5) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed) (N=11)
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with Dose Expansion Cohort: Ixazomib 4 mg (PI Naive) and is not related.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort: Ixazomib 4.0 mg (N=6) | Dose Escalation Cohort: Ixazomib 5.5 mg (N=5) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Naive) (N=5) | Dose Expansion Cohort: Ixazomib 4.0 mg (PI Exposed) (N=11)
Nausea (Gastrointestinal disorders) | 4 | 4 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 5
Fatigue (General disorders) | 2 | 3 | 3 | 6
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 2
Pyrexia (General disorders) | 1 | 1 | 1 | 5
Oedema peripheral (General disorders) | 3 | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 3 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 5
Hypotension (Vascular disorders) | 1 | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 1
Chills (General disorders) | 1 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Statistical Analysis Plan (2012-11-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT01318902/SAP_000.pdf
  • Study Protocol (2014-12-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT01318902/Prot_001.pdf